CLINICAL TRIAL: NCT06113042
Title: Effectiveness and Sustainability of a Community Child Health Model in Community Settings
Brief Title: KeySteps@JC Phase Two Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: KeySteps@JC 2.0
Record Dates: First submitted 2023-10-03; First posted 2023-11-02 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-08

CONDITIONS: Lifestyle Modification
Keywords: Community child health; Child development; Nutrition; Physical activity; Sleep; Healthy lifestyle; Lifestyle modification; KeySteps
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Comprehensive support (Group 1) (Experimental): Comprehensive health support will be performed both in district community hub and school. Interventional services include heath talks, learning packs, hub-based comprehensive lifestyle modification programme, school healthy environment evaluation.
  Interventions: Behavioral: Health talks, learning packs; Behavioral: Lifestyle modification programme; Behavioral: School healthy environment evaluation
- School-based support (Group 2) (Experimental): Interventional services will be performed in school only, including heath talks, learning packs, school-based lifestyle modification programme, school healthy environment evaluation.
  Interventions: Behavioral: Health talks, learning packs; Behavioral: Lifestyle modification programme; Behavioral: School healthy environment evaluation
- District-based support (Group 3) (Experimental): Interventional services will be performed in community hub only, including heath talks, learning packs, hub-based lifestyle modification programme.
  Interventions: Behavioral: Health talks, learning packs; Behavioral: Lifestyle modification programme
- Control (Group 4) (Placebo Comparator): Limited services will be provided including health talks and learning packs.
  Interventions: Behavioral: Health talks, learning packs

INTERVENTIONS:
Behavioral: Health talks, learning packs — All participants can join the health talks and receive the learning packs.
Behavioral: Lifestyle modification programme — In Group 1: The programme includes both knowledge and activity/practicum sessions for children and parents. It will be carried out in district community hubs.
  Group 2: The programme focuses on the knowledge sessions for parents. It will be carried out in schools.
  Group 3: The programme focuses on the activity/practicum sessions for children and parents. It will be carried out in district community hubs.
  Arms: Comprehensive support (Group 1); District-based support (Group 3); School-based support (Group 2)
Behavioral: School healthy environment evaluation — Evaluation on school healthy environment will be carried out in Group 1 and Group 2 to enhance the schools to provide a healthy school environment to children.
  Arms: Comprehensive support (Group 1); School-based support (Group 2)

SUMMARY:
This proposed 'KeySteps Phase Two Study' is a 5-year study, which aims to investigate the effectiveness and sustainability of a Community Child Health Model with different services related to healthy lifestyle programmes and health promotion implemented in community settings of deprived living areas. Potential participants are children studying or living in the five selected districts, namely Sham Shui Po, Yuen Long, Tuen Mun, Sha Tin and Kowloon City. Data including children's health and psychosocial conditions, and family demographics will be collected. In addition, subjects will receive on-site assessments on general health and development. Medical and health related events of subjects will be tracked through the existing health care system. Subjects will receive health promotion services and/or lifestyle modification programmes according to their needs.

DETAILED DESCRIPTION:
With the improved economy and rapid growth of socio-economic activities, the socioeconomic gaps between social groups in Hong Kong are widening continuously. According to the Hong Kong Poverty Report of Oxfam Hong Kong (OHK), the richest decile of households made 34.3 times more than the poorest decile prior the COVID pandemic (2019), that number surged to 47.3 times by the first quarter of 2022.1 Similar to the experience in other countries, children from low socio-economic status (SES) families in Hong Kong are at higher risk of physical health, psychological and behavioural problems including obesity/overweight and hypertension, visual, behavioural and learning problems.

Major chronic diseases such as central obesity, hypertension, diabetes mellitus, ischemic heart disease, degenerative retinal and other eye diseases are found to be rooted in childhood related to unhealthy lifestyles, adverse thriving and nutritional environment. The COVID-19 pandemic has exaggerated the existing risks and led to emerging threats among young children, especially in disadvantaged families in Hong Kong in the past two years. With the stringent social isolation, school suspension and home confinement, children's physical health, developmental and behavioral problems have worsened. Experience in a local project, KeySteps@JC funded by HKJC 2017-2022 showed that children in deprived districts were susceptible to nutritional imbalance, physical inactivity and weight problems, especially during the COVID-19 period. Another study also reported the overuse of electronic devices in disadvantaged families. Several other studies also indicated that there were adverse health effects related to COVID-19 pandemic including obesity, deteriorated physical fitness, visual impairment in particular myopia, sleep and emotional disturbance, decreased school readiness, and increased risk of child maltreatment, inattention/hyperactivity and neurodevelopmental disorders, etc.

Lifestyle modification addresses the poor lifestyle choices that are the root causes of chronic diseases. The goal of the lifestyle modification programme is to empower the patient with knowledge, skills, and a desire to create and maintain new habits which are needed to manage their chronic disease and potentially eliminate the root cause. Parental or family involvement in interventions is found to be impactful on lifestyle changes in children, leading to favourable health outcomes. As a result of modelling their parents' behaviour, children are more likely to adopt a healthy lifestyle if their parents demonstrate healthy lifestyle behaviours. Research also found that parents perceived social support to be a key enabler for children to eat healthfully and be active. Group-based health interventions may encourage the building of peer support with additional benefits of social support in the community.

Although lifestyle modification programmes seem promising to address the increasing need of young children, they have not been widely implemented in early childhood public health settings as a main health promotion and disease prevention strategy. This research is to investigate the effectiveness and sustainability of a Community Child Health Model with different services related to healthy lifestyle programmes and health promotion implemented in community settings of deprived living areas.

Potential participants are children studying or living in the five selected districts, namely Sham Shui Po, Yuen Long, Tuen Mun, Sha Tin and Kowloon City. Those districts shared some common disadvantaged backgrounds such as families with lower socio-economic status, mostly living in subdivided units and crowded housing, insufficient public play area and early childhood services. According to the Hong Kong Poverty Situation Report from Census and Statistics Department in 2018, Yuen Long ranked 2nd highest, Tuen Mun 4th, Sham Shui Po 5th, Sha Tin 6th and Kowloon City 9th in terms of 0-6 years old child living in poverty population.11 Moreover, Sham Shui Po was the second-highest district with subdivided units12and Kowloon City ranked third in terms of the number of partitioned flats and second-lowest districts in the public play space area managed by Leisure and Cultural Services Department (LCSD).

This study will be conducted in compliance with the protocol, Declaration of Helsinki and other applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Children are studying in kindergartens which agree to join the project.
2. Parent/legal guardian of the child consented the child's participation in to the study.
3. Participants of the Lifestyle modification Programme should be K1 students in academic year 2023/24 of the selected kindergartens and their parents/guardians.

Exclusion Criteria:

1. Parent/legal guardian of the child cannot understand Cantonese.
2. Parent/legal guardian of the child cannot read Chinese.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
weight | 5 years
  Assessing children's body weight (kg) to check for overweight or underweight.
Physical activity level | 5 years
  Assessing the physical activity intensity and duration (minutes) with the activity monitoring device (Actigraph).
Nutritional status | 5 years
  Assessing the nutritional status and dietary habits with the food frequency questionnaire (electronic version). The frequency and quantity of food intake will be recorded. The consumption of different kinds of nutrients will be calculated and compared with the reference levels to determine the adequacy.
Use of electronic devices | 5 years
  Assessing the duration of daily use of electronic devices.
Parental awareness | 5 years
  Assessing changes on parent's knowledge, attitudes and practices on child healthy lifestyle by a questionnaire. A 5-point scale is adopted. The higher the score, the better the result.

SECONDARY OUTCOMES:
Feedback evaluation | 5 years
  Obtaining the programme feedback from stakeholders on the project health service by a feedback questionnaire. A 6-point scale is adopted. The higher the score, the better the result.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick IP, MPH, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No